CLINICAL TRIAL: NCT07048509
Title: Difference in Acute Responses of Vascular Function to Moderate-intensity and High-intensity Interval Training in Healthy and Prehypertensive Individuals
Acronym: ACT-ON-ACUTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Simon Iskra, Principal Investigator, University of Ljubljana
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 0120-63/2025-2711-3; 802-15/2023-5 (Other Grant/Funding Number: University of Ljubljana (slo: Razvojni Sklad UL)); 005-1/2023 (Other Grant/Funding Number: University of Ljubljana (slo: Razvojni Sklad UL))
Record Dates: First submitted 2025-06-20; First posted 2025-07-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prehypertension (Elevated Blood Pressure) or Hypertension; Healthy
Keywords: aerobic exercise; vascular function; prehypertension
MeSH Terms: conditions — Prehypertension; Hypertension | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective double-blind crossover randomized study design
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normotensive (Placebo Comparator): Normotensives with ambulatory blood pressure measurements within the optimal range according to the 2023 ESH guidelines
  Interventions: Other: Control-no treatment; Other: Exercise
- Prehypertensive (Active Comparator): Prehypertensives with blood pressure within 120-139 mmHg systolic and/or 80-89 diastolic.
  Interventions: Other: Control-no treatment; Other: Exercise

INTERVENTIONS:
Other: Control-no treatment — 30 minutes of rest
Other: Exercise — 30 minutes of Moderate-Intensity Continuous Exercise
Other: Exercise — 30 minutes of High-Intensity Interval Exercise

SUMMARY:
In this study, the investigators will evaluate acute changes in vascular function measures after moderate-intensity continuous and high-intensity interval exercise in healthy and prehypertensive individuals. Participants will be subjected to three separate visits: control condition (30 min rest), moderate-intensity continuous exercise, and high-intensity interval exercise. The investigators will measure aerobic capacity using a cardiopulmonary exercise test (CPET) using indirect gas-exchange to derive subsequent exercise intensity and maximal oxygen uptake. The investigators will evaluate different measures of vascular function (Pulse-wave velocity, Flow-mediated slowing, microvascular function) before and after each condition.

The study will involve two groups of participants: healthy individuals and prehypertensive individuals. The investigators aim to establish the reliability and validity of less-established methods of vascular function assessment (flow-mediated slowing and microvascular function) against established measures (pulse-wave velocity). The acute response of vascular function to different exercise intensities has not yet been thoroughly researched using the aforementioned measures in individuals with similar characteristics to the proposed study cohort.

DETAILED DESCRIPTION:
This study is a work package of the ACT-ON project, aimed at establishing the reliability and validity of flow-mediated slowing and microvascular function, as well as determine the acute response of different vascular function measures to different exercise conditions. The investigators aimed to include vascular function measures evaluating different parts of the vasculature (e.g. central, peripheral and microvasculature) to establish whether the specific response differs between healthy participants and participants at risk of developing cardiovascular diseases.

Data collection will be conducted using a range of instruments and tools in the following order.

To ensure compliance with the inclusion criteria, participants will undergo a screening visit prior to the enrollment in the study. The visit will take place in the morning including the following assessments: Standardized blood pressure (M6, Omron, Japan), height (GPM, Model 101, Switzerland) and weight (InBody 720, Biospace, South Korea) measurement, as well as the administration of the GPAQ questionnaire. Female participants will additionally complete a Reproductive status Questionnaire (RSQ) (Schmalenberger & Eisenlohr-Moul, 2019) to determine eligibility based on previously established inclusion and exclusion criteria. Participants will be advised to refrain from physical activity, alcohol and caffeine consumption in the days leading up to the visit, as well as to arrive well rested and in a fasted state.

Study protocol

After enrollment in the study, participants will complete three visits with 72h between each visit. The visits will be completed at the same hour of the day to ensure minimal circadian variability. Participants will be advised to refrain from physical exercise and consumption of alcohol and caffeine in the days leading up to the first visit, as well as during the study. Additionally, they will be advised to arrive well rested and to consume a standardized meal 2-3 hours before the visit. To enable physical activity monitoring during the study, participants will wear wrist monitors with 24-h measurement of heart rate on the wrist (Vantage V3, Polar, Finland). In the event that physical activity is detected during the course of the study, participants will be excluded from the study. Additionally, participants will be required to maintain a dietary intake log during the duration of the study.

Body composition measurement using bioimpendance method (InBody 720, Biospace, South Korea) will be taken after arrival to the laboratory of the Institute of Sport, University of Ljubljana. After, participants will sit on a chair for 10 minutes in a quite environment with the hand extended and supinated, resting on a surface at heart level. Subsequently, three consecutive BP measurements will be taken using an automated upper-arm blood pressure monitor (M6, Omron, Japan) with one-minute intervals between each measurement. BP will be calculated as the average of the last two recordings.

Haemodynamics

Pulse Wave Velocity (PWV) Characteristics

The Vicorder device (software version 4; Skidmore Medical, United Kingdom) will be used to measure pulse wave characteristics (PWA) of the brachial artery and pulse wave velocity from the carotid to the femoral artery (cfPWV). This device uses an oscillometric technique to obtain the pulse wave. cfPWV measurements will be taken using a 10 cm cuff around the upper right thigh to detect the femoral pulse and a 3 cm cuff around the neck to detect the right carotid pulse. The neck cuff is designed to be positioned above one carotid artery, avoiding compression of the trachea and both carotid arteries simultaneously. The distance between the suprasternal notch and the cuff on the upper thigh will be measured according to the manufacturer's instructions. Both cuffs will automatically inflate simultaneously to 65 mmHg, with pulse waves recorded in 3 to 5 second intervals while the participant lies in a supine position.

Flow-Mediated Slowing (FMS)

The VICORDER® EndoCheck FMS model will be used for FMS determination. Testing will be conducted following the device instructions. The pulse wave velocity (PWV) on the upper arm was measured simultaneously between the wrist and upper part of the right arm over 10 minutes, with a 5-minute flow occlusion period. FMS will be determined by continuously measuring the minimal PWV compared to the baseline PWV, with the percentage change designated as FMS.

Microvascular function

Near-infrared spectroscopy (NIRS) will be used to assess microvascular function, using a sensor to determine relative changes in oxygenated (O2Hb) and deoxygenated (HHb) haemoglobin. The sensor will be placed on the anteromedial part of the forearm (flexor carpi radialis muscle), 2 cm below the medial epicondyle of the humerus. A continuous-wave NIRS system (PortaMon, Artinis, Netherlands) will be used. The sensor is equipped with six light sources operating at six wavelengths (759, 760, 763, 848, 844 in 848 nm) and an optode distance of 35 mm. The NIRS signal will be recorded at a sampling frequency of 10 Hz. Tissue Saturation Index (TSI) will be calculated based on the modified Beer-Lambert law using the following equation:

TSI= ([O2Hb])/(([HHb]+[O2Hb])) Microvascular function will be assessed concurrently with the FMS measurement. Based on changes of the TSI signal during and after the ischemic stimulus, several variables will be calculated to evaluate microvascular function.

Blood markers

Blood markers will be taken from the left median cubital vein by a licenced clinician following standardized protocol. A 7 mL sample will be taken before the start of vascular function measurements before and after each assigned condition. The analysis of the sample will include basic blood panel markers: total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), triglycerides, blood glucose.

Physical performance

To obtain physiological parameters, the investigators will use a gas analyzer CPET (COSMED, Italy). The device provides reliable values for oxygen uptake (VO2), carbon dioxide production (VCO2), and pulmonary ventilation (VE) on a breath-by-breath basis. Heart rate will be measured simultaneously with a heart rate monitor chest strap (Polar, model H10, Finland). Data will be recorded in 5-second intervals and automatically analyzed using the original Polar software.

Incremental cycling test

After 5 minutes of baseline measurements sitting on the stationary ergometer (Excalibur sport, Lode, Netherlands) the participants will begin warm-up for 5 minutes at 1 W/kg. After, the test will be performed, in a step-incremental protocol starting at 60 W and increase of 15 W/min every minute.

Exercise Interventions

Participants will undergo the following tests (with 72 hours between visits): a) 30 min of rest (control condition), followed by an incremental exercise test to determine maximal oxygen uptake and exercise intensity prescription based on ventilatory thresholds, and in a randomized fashion: b) An acute moderate-intensity training session, c) an acute high-intensity interval training session. All exercise stimuli will be performed on an electronically braked cycling ergometer. Exercise intensity will be individually adjusted based on exercise test results. The intensity and duration of exercise training sessions will be adjusted to achieve similar caloric expenditure. Participants will be advised to refrain from exercise, consummation of alcohol and caffeine in the days before and during the research period. Additionally, they will be instructed to arrive well rested and consume a standardized meal 2-3 hours before arriving for evaluation. All measurements will be conducted at the same time of day, between 8:00 and 12:00, to minimize circadian variability. Vascular function (PWV, FMS, NIRS, blood markers) will be assessed before the start and after the end of each exercise stimulus and control condition. Blood markers will be collected from the cubital vein before and immediately after exercise.

Participants will undertake 5 min of light-intensity warm-up. Moderate-intensity exercise will be performed as 30 minute of continuous cycling set to 65% of intensity at respiratory compensation point (RCP), which is used as a marker of maximal metabolic steady state during exercise. High-intensity exercise will be performed as 4 repetitions of 4-minute intervals at 95 - 100 % of RCP, with 3 minutes of passive rest. Heart rate will be used as an additional measure to ensure adherence to the correct intensity zone (Coates et al., 2023). During exercise, participants' O2Hb and HHb, as well as TSI response will be monitored using NIRS, along with heart rate and cycling load. To ensure minimal dispersion of the NIRS signal, the adipose tissue thickness (ATT) on the muscle belly of the measured muscles will be assessed and ATT measurements exceeding one half of the optode distance will be excluded. Blood pressure measurements will be taken upon arrival and after each interval, as well as immediately after cessation of exercise. Parameters during exercise will be used to determine the response to different exercise intensities.

ELIGIBILITY:
Inclusion Criteria:

Normotensive participants inclusion criteria:

* 18 - 50 years of age, BMI < 30, blood pressure (BP) within the optimal range according to the latest ESH guidelines (< 120 mmHg systolic and/or < 80 mmHg diastolic BP)
* Sedentary or low active according to the Global Physical Activity Questionnaire (GPAQ) (Armstrong & Bull, 2006; Lim et al., 2012)
* No prescribed medication and absence of chronic diseases

Inclusion criteria for prehypertensive individuals:

* 18 - 50 years of age, BMI < 30
* Diagnosed prehypertension by a clinican from the Hypertension clinic, University clinical centre of Ljubljana using established criteria
* Sedentary or low or moderately active according to the Global Physical Activity Questionnaire (GPAQ)
* No prescribed medication and absence of chronic diseases

Exclusion Criteria:

* Blood pressure out of the optimal range (normotensives)
* High level of phyisical activity (moderate or high active according to GPAQ)
* Hypotension
* Chronic diseases
* Prescribed medication
* Lower extremity injury in the last six months
* Menopause
* Absence of normal menstrual cycle
* Pregnancy
* Smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | At the beginning of each visit (T0) and immediately after each acute stimulus (T1)
  Arterial stiffness will be measured by pulse wave velocity
Microvascular function | At the beginning of each visit (T0) and immediately after each acute stimulus (T1)
  Microvascular function will be mesured using near-infrared spectroscopy during and after a 5-minute occlusion of the brachial artery.
Flow-mediated slowing | At the beginning of each visit (T0) and immediately after each acute stimulus (T1)
  Flow-mediated slowing will be measured by pulse wave velocity deceleration after occlusion of the brachial artery.

SECONDARY OUTCOMES:
Aerobic capacity | Baseline
  Aerobic capacity will be assessed using cardiopulmonary exercise test on a cycle ergometer.
Blood pressure | Baseline
  Systolic and Diastolic blood pressure will be measured using M6 Omron Device.
Blood markers | At the beginning of each visit (T0) and immediately after each acute stimulus (T1)
  Blood samples will be taken from the median cubital vein and will include basic blood panel markers (HDL-C, LDL-C, TC, TG, glucose...)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ljubljana, Faculty of sport, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon reasonable request.